CLINICAL TRIAL: NCT00653328
Title: A Phase II Study of Atrasentan (ABT-627) Plus DOXIL in Patients With Recurrent Ovarian, Fallopian Tube, or Peritoneal Serous Papillary Adenocarcinoma Following Platinum + Taxane Therapy
Brief Title: Ph II Atrasentan + DOXIL in Recurrent Ovarian/Fallopian/Peritoneal Serous Papillary Adenocarcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Abbott (drug manufacturer) discontinued manufacture of ABT-627
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Marta Crispens, MD, Associate Professor; Gynecological Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC GYN 0288; VU-VICC-GYN-0288 (Other: Vanderbilt-Ingram Cancer Center); VU-VICC-020947
Record Dates: First submitted 2008-04-03; First posted 2008-04-04 (Estimated); Results first posted 2011-04-21 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; fallopian tube cancer; peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Atrasentan; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Therapeutic Intervention (Experimental)
  Interventions: Drug: atrasentan hydrochloride; Drug: doxil

INTERVENTIONS:
Drug: atrasentan hydrochloride — Atrasentan 10 mg orally everyday continuously beginning on Day 1.
  Other Names: ABT-627; Xinlay
Drug: doxil — 50 mg/m2 intravenously every 28 days
  Other Names: pegylated liposomal doxorubicin hydrochloride (Doxil)

SUMMARY:
RATIONALE: There is emerging data to suggest that the optimal use of angiogenesis inhibitors may be in combination with chemotherapy. The optimal use of atrasentan may be in combination with chemotherapy in women with relapsed and refractory ovarian cancer,fallopian tube cancer, and peritoneal serous papillary adenocarcinoma. Due to its manageable toxicity profile, ease of administration, and activity in both platinum sensitive as well as platinum-resistant patients, Doxil has become the 2nd-line treatment of choice for women with advanced stage ovarian cancer that has progressed following 1st-line platinum/taxane therapy.

PURPOSE: To determine if a treatment combination of atrasentan + Doxil is an effective 2nd line treatment in patients with recurrent ovarian cancer, fallopian tube cancer, or peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the median time to tumor progression in patients with recurrent ovarian epithelial cancer, fallopian tube adenocarcinoma, or peritoneal serous papillary adenocarcinoma treated with Doxil and atrasentan hydrochloride.

Secondary

* To determine the objective response rate and survival of patients treated with this regimen.
* To determine the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to response to prior treatment with platinum-taxane (sensitive vs resistant).

Patients will be administered Doxil 50 mg/m2 intravenous every 28 days and take atrasentan 10 mg orally everyday continuously beginning on Day 1. Patients will continue Doxil + atrasentan in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 30 days and every 2 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma arising from the ovary, fallopian tubes, or peritoneum (i.e., peritoneal serous papillary adenocarcinoma)
* Received prior treatment with either cisplatin or carboplatin in combination with paclitaxel or docetaxel as first-line chemotherapy
* Radiographic evidence of progressive disease and/or a doubling of CA-125 levels ≥ 70 IU/mL following first-line chemotherapy
* Measurable disease as defined by RECIST criteria
* No CNS metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Absolute neutrophil count ≥ 1,500/μL
* Hemoglobin ≥ 9.5 g/dL
* Platelets > 100,000/μL
* Serum creatinine ≤ 1.5 times upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 times ULN
* AST and ALT ≤ 2.5 times ULN (≤ 5.0 times ULN if liver metastases are present)
* LVEF ≥ 50% by MUGA
* Not pregnant or nursing
* Negative pregnancy test
* Surgically sterile or must use effective contraception
* No known HIV positivity or AIDS
* No uncontrolled heart disease, diabetes, or other medical condition that would place the patient at unacceptably high risk for toxicity
* No New York Heart Association class I-IV heart failure

Exclusion Criteria:

Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from all prior toxicities to ≤ grade 1 by NCI-CTC Version 2 criteria
* No other prior systemic therapies for this cancer except cisplatin or carboplatin in combination with paclitaxel or docetaxel as first-line chemotherapy
* More than 4 weeks since prior chemotherapy
* No concurrent anticancer therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2003-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marta Crispens, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (6):
- United States (6):
  - Central Georgia Hematology Oncology Associates, P.C., Macon, Georgia
  - Kentuckiana Cancer Institute, Louisville, Kentucky
  - The Jones Clinic, Germantown, Tennessee
  - Jackson-Madison County Hospital, Jackson, Tennessee
  - St. Thomas Health Services, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period = 5/28/2003 through 9/15/2006
Pre-assignment Details: A total of 16 people signed consent to take part in this study; of those, one withdrew consent before beginning treatment.
Groups:
- Altrasentan + Doxil: Atrasentan, 10 mg orally everyday continuously beginning on Day 1. Doxil. 50 mg/m2 intravenously every 28 days
Period: Overall Study
Arm/Group | Altrasentan + Doxil
Started | 15
Completed | 0
Not Completed | 15
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 2
Not completed — Disease progression | 10
Not completed — Drug manufacturer no longing making drug | 2

BASELINE CHARACTERISTICS:
Arm/Group | Altrasentan + Doxil
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 8
Age Continuous [Mean (Standard Deviation); unit: years] | 66 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Median Time to Tumor Progression
Description: Tumor progression is determined by appropriate imaging techniques according to RECIST criteria or by CA-125 serum level >=2x baseline and >=70 IU/ml, confirmed by a second determination at least 28 days after the first determination
Time Frame: Date on study to the date of measured progressive disease, every 2 cycles (2 months)
Population: Patients available for measurement of tumor response. One patient withdrew after beginning treatment.
Measure: Median (Full Range); unit: Months
Arm/Group | Altrasentan + Doxil
Number analyzed (Participants) | 14
Months | 1 (2.9) [0 to 11]

2. Secondary Outcome: Number of Patients With Objective Response
Description: Patient response to treatment:
  Progressive disease (PD): >=20% increase in sum of longest diameter (LD) of target lesion(s), taking as reference smallest sum LD recorded since treatment started, or appearance of >= 1 new lesions, and/or 2x CA-125 levels to >=70 IU/ml, confirmed by second measurement after 28 days Complete response (CR): disappearance of all target lesions Partial response (PR): >=30% decrease in sum of LD of target lesion(s), taking as reference baseline sum LD Stable disease (SD): neither sufficient shrinkage to qualify as PR nor sufficient increase to qualify as PD
Time Frame: At month 2 and monthly thereafter to cessation of treatment
Population: Patients who were available for measurement of tumor response.One patient withdrew after beginning treatment and was not available for measurement.
Measure: Number; unit: participants
Arm/Group | Altrasentan + Doxil
Number analyzed (Participants) | 14
participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 3
  Progressive Disease | 11

3. Secondary Outcome: Overall Survival
Time Frame: Date on study to date of death from any cause
Population: All patients who received treatment. Two patients alive at last follow-up.
Measure: Median (Full Range); unit: Months
Arm/Group | Altrasentan + Doxil
Number analyzed (Participants) | 13
Months | 10 [1 to 33]

4. Secondary Outcome: Number of Patients With Worst Grade Toxicities
Description: Not all participants necessarily have an adverse event, thus not everyone will be accounted for in worst-grade toxicities. Likewise, one participant can potentially have more than one event in various grades 1-5 which accounts for the difference in number of patients analyzed and total number in the worst-grade toxicity tables. Tables represent the number of patients with worst-grade toxicity at each of five grades (grade 1, least severe; to grade 5, most severe) following NCI Common Toxicity Criteria
Time Frame: Weekly for 2 weeks, then monthly for 5 months
Measure: Number; unit: participants
Arm/Group | Altrasentan + Doxil
Number analyzed (Participants) | 15
participants
  Number of participants with worst grade toxicity 1 | 5
  Number of participants with worst grade toxicity 2 | 3
  Number of participants with worst grade toxicity 3 | 3
  Number of participants with worst grade toxicity 4 | 0
  Number of participants with worst grade toxicity 5 | 0

ADVERSE EVENTS:
Arm/Group | Altrasentan + Doxil
Serious Adverse Events (participants affected / at risk) | 5/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Altrasentan + Doxil (N=15)
Pericardial effusion (Cardiac disorders) | 1 (1)
Thromboembolism (Vascular disorders) | 1 (1)
Fatigue (General disorders) | 3 (5)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Death (General disorders) | 1 (1)
edema (General disorders) | 1 (2)
fever (General disorders) | 2 (2)
fatigue (General disorders) | 2 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2)
pelvic pain (Reproductive system and breast disorders) | 1 (1)
urinary frequency (Renal and urinary disorders) | 1 (1)
hemoglobin (Investigations) | 2 (2)
abdominal cramping (Gastrointestinal disorders) | 1 (1)
hot flashes (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Altrasentan + Doxil (N=15)
Hemoglobin (Blood and lymphatic system disorders) | 7 (50)
fatigue (General disorders) | 10 (34)
Hypoalbuminemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2)
pelvic pain (Reproductive system and breast disorders) | 2 (2)
Urinary urgency (Renal and urinary disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 5 (8)
Vomiting (Gastrointestinal disorders) | 4 (5)
Abdominal Pain (Gastrointestinal disorders) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (11)
Hot flashes (Vascular disorders) | 2 (2)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Leukocytes (Blood and lymphatic system disorders) | 4 (29)
neutrophils, granulocytes (Investigations) | 2 (25)
platelets (Investigations) | 1 (14)
arrhythmias (Cardiac disorders) | 1 (1)
edema (General disorders) | 8 (13)
hypotension (Vascular disorders) | 2 (2)
fever (General disorders) | 2 (2)
rigors, chills (General disorders) | 1 (1)
sweating (Vascular disorders) | 1 (1)
weight gain (Investigations) | 4 (4)
alopecia (Skin and subcutaneous tissue disorders) | 4 (11)
bruising (Injury, poisoning and procedural complications) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 3 (8)
infectious wound (Infections and infestations) | 1 (2)
endrocrine (Endocrine disorders) | 1 (1)
anorexia (Psychiatric disorders) | 2 (3)
constipation (Gastrointestinal disorders) | 6 (8)
dehydration (Gastrointestinal disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 2 (2)
dysphagia (Gastrointestinal disorders) | 2 (2)
GI other (Gastrointestinal disorders) | 7 (12)
mouth dryness (Gastrointestinal disorders) | 1 (1)
hemorrhage (General disorders) | 1 (1)
alkaline phosphatase (Investigations) | 2 (2)
SGOT (Hepatobiliary disorders) | 2 (5)
SGPT (Hepatobiliary disorders) | 2 (3)
infection without neutropenia (Infections and infestations) | 2 (2)
hyperglycemia (Metabolism and nutrition disorders) | 5 (11)
hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
hypokalemia (Metabolism and nutrition disorders) | 1 (2)
metabolic, other (Metabolism and nutrition disorders) | 3 (5)
arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
dizziness (Nervous system disorders) | 1 (1)
insomnia (Psychiatric disorders) | 3 (7)
mood alteration (Psychiatric disorders) | 4 (6)
neuropathy (Nervous system disorders) | 7 (12)
dry eye (Eye disorders) | 2 (3)
tearing (Eye disorders) | 1 (2)
arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2)
headache (Nervous system disorders) | 4 (7)
chest pain (Cardiac disorders) | 1 (1)
neck pain (Musculoskeletal and connective tissue disorders) | 1 (12)
pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pulmonary, other (Respiratory, thoracic and mediastinal disorders) | 2 (2)
creatinine (Investigations) | 2 (2)
dysuria (Renal and urinary disorders) | 2 (2)
Renal, other (Renal and urinary disorders) | 2 (2)
constitutional symptoms (General disorders) | 1 (1)
pain (Musculoskeletal and connective tissue disorders) | 2 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes